CLINICAL TRIAL: NCT01179672
Title: Treatment of Patients With Diabetic Peripheral Neuropathic Pain in China: Duloxetine Versus Placebo
Brief Title: A Study in Participants With Diabetic Peripheral Neuropathic Pain in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13649; F1J-MC-HMGV (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Diabetic Neuropathy, Painful
Keywords: Diabetic Peripheral Neuropathic Pain
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — 30 mg administered orally (po), QD for 1 week; 60 mg administered po, QD for remaining 11 weeks; 30 mg administered po, QD for 1 week during taper period
  Other Names: Cymbalta; LY248686
  Arms: Duloxetine
Drug: Placebo — Administered po, QD for 12 weeks; administered po, QD for 1 week during taper period
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess the efficacy of duloxetine 60 milligrams (mg) once daily (QD) compared with placebo, on the change in pain severity from baseline to 12 weeks as measured by the weekly mean of the daily pain scores recorded in the participant's diary in participants with diabetic peripheral neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Present with pain due to bilateral peripheral neuropathy

  * Participants must have pain caused by Type 1 or Type 2 diabetes mellitus
  * Pain must begin in the feet with relatively symmetrical onset
  * Daily pain should be present for at least 6 months
  * Diagnosis must be confirmed by a score of at least 3 on the Michigan Neuropathy Screening Inventory (MNSI)
* Females must test negative for a serum pregnancy test at Screening. Females of child-bearing potential (who are not surgically sterilized and between menarche and 1 year postmenopause) must agree to use a medically acceptable and reliable means of birth control, during the study and for 1 month following the last study dose.
* Stable glycemic control as assessed by a physician investigator and a glycosylated hemoglobin (HbA1c) <12% before randomization
* Score of greater than or equal to 4 on the Brief Pain Inventory (BPI) 24-hour average pain item at Screening.
* Full completion of the daily diaries for at least 80% of the days between the second and third time you come to the hospital (Screening).

Exclusion Criteria:

* Currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Current (less than or equal to 1 year) Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) Axis I diagnosis of major depressive disorder, dysthymia, anxiety disorders (excluding phobias), alcohol or eating disorders as determined by the Mini-International Neuropsychiatric Interview (MINI) or a previous diagnosis
* DSM-IV diagnosis of mania, bipolar disorder, or psychosis determined either by participant history or by diagnosis using specific MNSI modules
* Serious or unstable cardiovascular, hepatic, renal, respiratory, or hematologic illness, symptomatic peripheral vascular disease, or other medical condition or psychological conditions that in the opinion of investigator would compromise participation or be likely to lead to hospitalization during the course of the study.
* At Screening alanine transaminase (ALT) greater than 2 times upper limit of normal (ULN), based on central laboratory reference ranges times ULN, based on central laboratory reference ranges
* Prior renal transplant, current renal dialysis, or serum creatinine laboratory value >1.5 times ULN, based on central laboratory reference ranges at Screening.
* Historical exposure to drugs known to cause neuropathy, or a history of a medical condition, including pernicious anemia and hypothyroidism, that could have been responsible for neuropathy
* Pain that cannot be clearly differentiated from or conditions that interfere with the assessment of the diabetic neuropathy pain. Examples of painful conditions that could be confused with diabetic neuropathy pain include peripheral vascular disease, neurological disorders unrelated to diabetic neuropathy, skin condition in the area of the neuropathy that could alter sensation, other painful conditions
* Participants who have previously completed or withdrawn from this study or have been previously treated with duloxetine, including participants who participated in study F1J-MC-HMEQ (NCT00408993), even those in the placebo arm
* Participants taking excluded medications that cannot be stopped at Screening
* Treatment with a monoamine oxidase inhibitor (MAOI) or fluoxetine within 30 days of the third Screening
* Participants with a positive Hepatitis B surface antigen and/or Hepatitis C antibody are to be excluded if they have any of the following:

  * Hepatic dysfunction as determined by the investigator or
  * Clinical manifestations of liver disease within the previous year such as unexplained pruritus, unexplained dark urine, jaundice, unexplained right upper quadrant tenderness, unexplained "flu-like" symptoms or
  * Aspartate transaminase (AST), ALT, or bilirubin above the normal reference range.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- China (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bengbu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changchun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chengdu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chongqing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jinan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Qingdao
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shantou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shijiazhuang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tianjin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xi'an
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yueyang

REFERENCES:
- [Derived] Gao Y, Guo X, Han P, Li Q, Yang G, Qu S, Yue L, Wang CN, Skljarevski V, Duenas H, Raskin J, Gu L. Treatment of patients with diabetic peripheral neuropathic pain in China: a double-blind randomised trial of duloxetine vs. placebo. Int J Clin Pract. 2015 Sep;69(9):957-66. doi: 10.1111/ijcp.12641. Epub 2015 May 4. PMID 25939897

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants tapered off study drug after either completing the 12 weeks of treatment or discontinued treatment early.
Groups:
- Duloxetine: 30 milligrams (mg) duloxetine capsule administered orally, once daily (QD) during Week 1 then 60 mg duloxetine capsule orally, QD for the remaining 11 weeks of treatment. After a total 12 weeks of treatment or early discontinuation participants tapered off study drug (30 mg duloxetine capsule QD) for 1 week during taper.
- Placebo: Placebo administered orally, QD for 12 weeks of the treatment and orally, QD for 1 week during taper.
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 203 | 202
Received at Least 1 Dose of Study Drug | 202 | 202
Entered Taper | 181 | 177
Completed | 173 | 176
Not Completed | 30 | 26
Not completed — Adverse Event | 17 | 8
Not completed — Withdrawal by Subject | 10 | 12
Not completed — Entry Criteria Not Met | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Duloxetine: 30 mg duloxetine capsule administered orally, QD during Week 1 then 60 mg duloxetine capsule orally, QD for remaining 11 weeks of the treatment. After a total 12 weeks of treatment or early discontinuation, participants tapered off study drug (30 mg duloxetine capsule orally, QD) for 1 week during taper.
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 203 | 202 | 405
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.56 (9.65) | 61.17 (9.42) | 61.37 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 111 | 223
  Male | 91 | 91 | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 203 | 202 | 405
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 203 | 202 | 405
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 203 | 202 | 405
Diabetes Disease Characteristics-Types of Diabetes [Number; unit: participants]
  Type I Diabetes | 3 | 3 | 6
  Type II Diabetes | 200 | 199 | 399
Diabetes Disease Characteristics [Mean (Standard Deviation); unit: years]
  Duration of Diabetes | 11.53 (6.81) | 11.38 (7.47) | 11.45 (7.14)
  Duration of Diabetic Neuropathy | 3.47 (3.91) | 3.07 (3.13) | 3.27 (3.55)
  Duration of Diabetic Neuropathy Pain | 3.06 (3.70) | 2.59 (2.69) | 2.83 (3.24)
Weekly Mean of 24-Hour Average Pain [Mean (Standard Deviation); unit: units on a scale] — Participants measured their pain on an 11-point Likert scale that was completed daily. The scale ranged from 0 (no pain) to 10 (worst possible pain). The participant-recorded average pain due to diabetic neuropathy over the previous 24 hours.
  units on a scale | 5.72 (1.72) | 5.62 (1.66) | 5.67 (1.69)
Brief Pain Inventory (BPI)-Severity Average Pain in the Last Week [Mean (Standard Deviation); unit: units on a scale] — BPI-Severity Modified Short Form Severity was a self-reported scale that measured the severity of pain. Severity scores ranged from 0 (no pain) to 10 (pain as bad as you could imagine). There were 4 questions assessing the severity for worst pain, least pain, average pain, and the pain right now.
  units on a scale | 5.97 (1.70) | 5.86 (1.64) | 5.91 (1.67)
Clinical Global Impression of Severity (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — Number of participants analyzed was: Duloxetine treatment =126 and Placebo=136. Data from 9 sites were not included in baseline analysis due to wrong questionnaire used. CSI-S was administered by the investigator in the presence of the participant and measured severity of illness at baseline with scores ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
  units on a scale | 4.76 (1.22) | 4.66 (1.07) | 4.71 (1.14)
Short Form-McGill Pain Questionnaire (SF-MPQ), Sensory Portion Total Score [Mean (Standard Deviation); unit: units on a scale] — SF-MPQ sensory portion was a self-reported instrument consisting of 11 sensory descriptors describing pain, each rated on an intensity scale from 0 (none) to 3 (severe). Total scores ranged from 0 to 33.
  units on a scale | 12.24 (6.39) | 11.81 (5.52) | 12.02 (5.97)
BPI-Interference Average Score [Mean (Standard Deviation); unit: units on a scale] — BPI-Interference Score was self-reported scale that measured interference of pain based on the average of the 7 questions assessing the interference of pain for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The average interference scores ranged from 0 (does not interfere) to 10 (completely interferes).
  units on a scale | 4.38 (2.29) | 4.08 (2.30) | 4.23 (2.30)
Sheehan Disability Scale (SDS) Total Score [Mean (Standard Deviation); unit: units on a scale] — SDS was self-reported and used to assess the effect of the participant's symptoms on their work (Item 1), social life (Item 2), and family life (Item 3). Each item was measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. SDS Total Score was the sum of the 3 items and ranged from 0 to 30 with higher values indicating greater disruption in the participant's work/social/family life. Scores ≥5 were associated with significant functional impairment.
  units on a scale | 11.16 (7.59) | 10.54 (7.31) | 10.85 (7.45)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline at 12-Week Endpoint in the Weekly Mean of Pain Severity Score
Description: 24-hour average pain severity scores were recorded daily by the participant on an 11-point Likert scale, an ordinal scale, with scores ranging from 0 (no pain) to 10 (worst possible pain). The weekly mean was calculated. A negative change indicated an improvement in participant's condition. Least squares (LS) mean was calculated using mixed model repeating measures (MMRM) and adjusted for treatment, pooled investigator, visit, and treatment-by-visit interaction, as well as baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, 12 weeks
Population: Intent-to-treat (ITT) principle was applied: All participants with a baseline and 12-week 24-hour average pain score based on the randomized group were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine: 30 mg duloxetine capsule administered orally, QD during Week 1, then 60 mg duloxetine capsule orally QD for remaining 11 weeks of the treatment. After a total 12 weeks of treatment or early discontinuation, participants tapered off study drug (30 mg duloxetine capsule orally, QD) for 1 week during taper.
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 172 | 173
units on a scale | -2.40 (0.14) | -1.97 (0.14)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.82 to -0.04]

2. Secondary Outcome: Mean Change From Baseline at 12-Week Endpoint in Weekly Mean of Night Pain and Worst Pain
Description: 24-hour average night pain and worst pain severity scores were recorded daily on an 11-point Likert scale, an ordinal scale, with scores ranging from 0 (no pain) to 10 (worst possible pain). A negative change indicated an improvement in the participant's condition. LS mean was calculated using MMRM and adjusted for treatment, pooled investigator, visit, and treatment-by-visit interaction, as well as the baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, 12 weeks
Population: ITT principle was applied: All participants with a baseline and 12-week 24-hour night pain score and worst pain score based on the randomized group were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Duloxetine: 30 mg duloxetine capsule administered orally, QD during Week 1, then 60 mg duloxetine capsule orally, QD for remaining 11 weeks of the treatment. After a total 12 weeks of treatment or early discontinuation, participants tapered off study drug (30 mg duloxetine capsule orally, QD) for 1 week during taper.
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 172 | 173
units on a scale
  Night Pain | -2.65 (0.15) | -2.11 (0.15)
  Worst Pain | -2.80 (0.16) | -2.25 (0.17)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — P-value is for mean change from baseline to 12-week endpoint in night pain; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.95 to -0.14]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.017, Mixed Models Analysis — P-value is for mean change from baseline to 12 week endpoint in worst pain; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-1.00 to -0.10]

3. Secondary Outcome: Mean Change From Baseline at 12-Week Endpoint in the BPI-Severity Scale
Description: BPI-Severity Scale was a self-reported scale that measured the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). A negative change indicated an improvement in the participant's condition. LS mean was calculated using MMRM and adjusted for treatment, pooled investigator, visit, and treatment-by-visit interaction, as well as baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, 12 weeks
Population: ITT principle was applied: All participants with a baseline and 12-week, 24-hour BPI-Severity score based on the randomized group were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 175 | 173
units on a scale | -2.50 (0.15) | -2.00 (0.15)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.016, Mixed Models Analysis; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.90 to -0.09]

4. Secondary Outcome: Mean Change From Baseline at 12-Week Endpoint in the CGI-S Scale
Description: CGI-S was administered by the investigator in the presence of the participant and measured the severity of illness at the time of assessment compared with start of treatment; CGI-S scores ranged from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). A negative change indicated an improvement in the participant's condition. LS mean was calculated using MMRM and adjusted for treatment, pooled investigator, visit, and treatment-by-visit interaction, as well as baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, 12 weeks
Population: ITT principle was applied: All participants with a baseline and 12-week CGI-S score based on the randomized group were analyzed. Data from 9 sites was not included in analysis due to wrong questionnaire used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 108 | 118
units on a scale | -1.40 (0.10) | -1.17 (0.10)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.081, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.48 to 0.03]

5. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Scale at 12-Week Endpoint
Description: PGI-I was self-reported and measured a participant's perception of improvement at the time of assessment compared with the start of treatment. Scores ranged from 1 (very much better) to 7 (very much worse). LS mean was calculated using MMRM and adjusted for treatment, pooled investigator, visit, and treatment-by-visit interaction, as well as baseline score and baseline score-by-visit interaction.
Time Frame: 12 weeks
Population: All participants with a baseline and 12-week PGI-I score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 173 | 176
units on a scale | 2.44 (0.07) | 2.65 (0.07)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.034, Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.40 to -0.02]

6. Secondary Outcome: Mean Change From Baseline at 12-Week Endpoint in the Sensory Subscale of the SF-MPQ
Description: SF-MPQ was a self-reported instrument that consisted of 11 sensory descriptors describing pain. The descriptors were rated on an intensity scale from 0 (none), 1 (mild), 2 (moderate) or 3 (severe). Three (3) pain scores were derived from the sum of the intensity rank values of the words chosen for sensory descriptors. The SF-MPQ sensory subscale was the sum of the 11 scores (ranged from 0 to 33, with 33 being the worst pain). A negative change indicates an improvement. LS mean was calculated using analysis of covariance (ANCOVA) adjusted for treatment, pooled investigator and baseline.
Time Frame: Baseline, 12 weeks
Population: ITT principle was applied: All participants with a baseline and 12 weeks SF-MPQ score based on the randomized group were analyzed; last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 188 | 180
units on a scale | -6.45 (0.36) | -5.33 (0.39)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.022, ANCOVA; ANCOVA adjusted for treatment, pooled investigator and baseline; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-2.07 to -0.16]

7. Secondary Outcome: Percentage of Participants Who Experience Equal to or Greater Than 30%, 50% or 75% Reduction From Baseline at 12-Week Endpoint in Weekly Mean of Average Daily Pain
Description: 24-hour self-assessment of average daily pain was recorded in the participants diary based on an 11 point Likert scale with scores ranging from 0 (no pain) to 10 (worst possible pain). Percentage of participants was calculated as: (number of participants with 30% [or 50% or 75%] reduction in average daily pain) divided by (number of participants) multiplied by 100.
Time Frame: Baseline, 12 weeks
Population: All participants with a baseline and postbaseline 24-hour average pain score.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 200 | 198
percentage of participants
  ≥30% Reduction | 61.5 | 49.0
  ≥50% Reduction | 42.0 | 28.8
  ≥75% Reduction | 14.5 | 9.6
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.014, Cochran-Mantel-Haenszel — P-value is for ≥30% reduction in 24-hour average pain; Cochran-Mantel-Haenszel test was stratified by pooled investigator
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — P-value is for ≥50% reduction in 24-hour average pain; Cochran-Mantel-Haenszel test was stratified by pooled investigator
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.193, Cochran-Mantel-Haenszel — P-value is for ≥75% reduction in 24-hour average pain; Cochran-Mantel-Haenszel test was stratified by pooled investigator

8. Secondary Outcome: Percentage of Participants Who Experienced Equal to or Greater Than 30%, 50% or 75% Reduction From Baseline at 12-week Endpoint in BPI-Severity Average Pain Score
Description: BPI-Severity scale was a self-reported scale that measured the severity of pain based on the average pain experienced over the past 24 hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). A negative change indicated an improvement in the participant's condition. Percentage of participants was calculated as: (number of participants with 30% [or 50% or 75%] reduction in BPI-Severity average pain) divided by (number of participants) multiplied by 100.
Time Frame: Baseline, 12 weeks
Population: All participants with a baseline and postbaseline BPI-Severity average pain scores.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 200 | 197
percentage of participants
  ≥30% Reduction | 63.0 | 46.7
  ≥50% Reduction | 46.0 | 29.4
  ≥75% Reduction | 15.0 | 9.6
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — P-value is for ≥30% reduction in 24-hour BPI-Severity average pain; Cochran-Mantel-Haenszel test was stratified by pooled investigator
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — P-value is for ≥50% reduction in 24-hour BPI-Severity average pain; Cochran-Mantel-Haenszel test was stratified by pooled investigator
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.168, Cochran-Mantel-Haenszel — P-value is for ≥75% reduction in 24-hour BPI-Severity average pain; Cochran Mantel Haenszel test was stratified by pooled investigator

9. Secondary Outcome: Mean Change From Baseline at 12-week Endpoint in the BPI Interference Score
Description: BPI-Interference Score was a self-reported scale that measured the interference of pain based on the average of the 7 questions assessing the interference of pain for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The average interference scores ranged from 0 (does not interfere) to 10 (completely interferes). A negative change indicates an improvement in the participant's condition. LS means was calculated using MMRM and adjusted treatment, pooled investigator, visit, and treatment-by-visit interaction, baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, 12 weeks
Population: All participants with non-missing BPI-Interference score at baseline and 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 173 | 176
units on a scale | -2.42 (0.13) | -1.82 (0.14)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-0.96 to -0.24]

10. Secondary Outcome: Mean Change From Baseline at 12 Week Endpoint in the SDS Total Score
Description: SDS was self-reported and used to assess the effect of the participant's symptoms on their work (Item 1), social life (Item 2), and family life (Item 3). Each item was measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. SDS total score was the sum of the 3 items and ranged from 0 to 30, with higher values indicating greater disruption in the participant's work/social/family life. Scores ≥5 were associated with significant functional impairment. A negative change indicated an improvement in the participant's condition. LS mean was adjusted using MMRM and adjusted for treatment, pooled investigator, visit, and treatment-by-visit interaction, baseline score and baseline score-by-visit interaction.
Time Frame: Baseline, 12 weeks
Population: All participants with non-missing SDS Total Score at baseline and 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 172 | 175
units on a scale | -6.36 (0.40) | -5.09 (0.42)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.020, Mixed Models Analysis; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-2.33 to -0.20]

ADVERSE EVENTS:
Groups:
- Duloxetine Treatment: 30 mg duloxetine capsule administered orally, QD during Week 1 of the treatment; 60 mg capsule administered orally, QD for remaining 11 weeks of the treatment;
- Placebo Treatment: Placebo administered orally, QD for 12 weeks of the treatment.
- Duloxetine Taper: After 12 weeks of treatment or early discontinuation, 30 mg duloxetine capsule administered orally, QD for 1 week during taper.
- Placebo Taper: After 12 weeks of treatment or early discontinuation, placebo administered orally, QD for 1 week during taper.
Arm/Group | Duloxetine Treatment | Placebo Treatment | Duloxetine Taper | Placebo Taper
Serious Adverse Events (participants affected / at risk) | 4/202 | 3/202 | 3/181 | 1/177
Other Adverse Events (participants affected / at risk) | 93/202 | 71/202 | 8/181 | 5/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine Treatment (N=202) | Placebo Treatment (N=202) | Duloxetine Taper (N=181) | Placebo Taper (N=177)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Duloxetine Treatment (N=202) | Placebo Treatment (N=202) | Duloxetine Taper (N=181) | Placebo Taper (N=177)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Amaurosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (10) | 4 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 21 (23) | 7 (7) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 9 (10) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 10 (10) | 4 (6) | 0 (0) | 0 (0)
Hunger (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Sluggishness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatty liver alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord injury cauda equina (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11) | 8 (8) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 (9) | 5 (5) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic autonomic neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 17 (18) | 9 (9) | 0 (0) | 0 (0)
Dreamy state (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Formication (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 3 (4) | 1 (1) | 1 (1)
Hypersomnia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 17 (18) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphoria (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fear (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food aversion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Illusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Mutism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tic (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/91 (1) | 0/91 (0) | 0/85 (0) | 0/76 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days